CLINICAL TRIAL: NCT01931774
Title: Is Acne a Skin Disease Affecting the Brain Functions? Neurocognition in Patients With Acne Vulgaris
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Erdem Deveci, Ass.Prof., Bezmialem Vakif University
Other Study IDs: Etik Kurul Karar No:36/14
Record Dates: First submitted 2013-08-27; First posted 2013-08-29 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris cognitive functions
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acne Patients
- Control Subjects: From General Population

SUMMARY:
Acne vulgaris usually causes psychological distress, depression, and anxiety disorders that may impair neurocognitive functions such as memory, attention, psychomotor speed, and executive functions, which are also common psychiatric disorders in patients with acne.

The purpose of this study is to determine cognitive functioning in treatment naive acne patients, without a history of any psychiatric disorder.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

The participants that had a symptom or a history of mental retardation (IQ < 70), serious head trauma, seizures or any other mental disorder, and participants on any medical treatment will be excluded. Participants with a family history (first degree relatives) of schizophrenia, bipolar disorder or schizoaffective disorder will also be excluded to avoid the negative effect of these disorders on cognitive functions. The same exclusion criteria will also be applied to the control group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acne patients referred to the dermatology outpatient clinic of our university and healthy controls matched with the patient group for age, gender and years of education. Controls will be taken from the general population
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Cognitive functions | baseline

SECONDARY OUTCOMES:
anxiety | baseline

OTHER OUTCOMES:
depression | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Erdem Deveci, Ass.Prof., Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University Hospital, Istanbul, Turkey (Türkiye)